CLINICAL TRIAL: NCT02865460
Title: A Randomized, Double-blind Placebo-controlled Phase III Trial of Coenzyme Q10 in Gulf War Illness
Brief Title: Coenzyme Q10 Phase III Trial in Gulf War Illness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLD-04-15F
Record Dates: First submitted 2016-07-28; First posted 2016-08-12 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Gulf War Illness; Chronic Fatigue; Ubiquinol; Coenzyme Q10
Keywords: Chronic Pain; Cognitive Disorders; Inflammation; Neurologic manifestations; Dementia; Mental Disorders; Ubiquinol/ubiquinone; Pathologic Processes; Nervous System Diseases; Hormones, Hormone Substitutes, and Hormone Antagon; Anti-Inflammatory Agents; Pharmacologic Actions; Therapeutic Uses; Physiological Effects of Drugs; Gulf war illness; Chronic fatigue
MeSH Terms: conditions — Chronic Pain; Cognitive Dysfunction; Inflammation; Neurologic Manifestations; Dementia; Mental Disorders; Pathologic Processes; Nervous System Diseases | interventions — ubiquinol; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ubiquinol (Experimental): Take oral tablets as directed (2x200 mg for 2 months; 1x200 mg for 4 months) with food each morning- upon waking
  Interventions: Drug: Ubiquinol
- Placebo (Placebo Comparator): Take oral tablets as directed (2x200 mg for 2 months; 1x 200 mg for 4 months) with food each morning-upon waking
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ubiquinol — Take oral tablets as directed (2x200 mg for 2 months; 1x200 mg for 4 months) with food each morning- upon waking
  Other Names: Coenzyme Q10, CoQ10
  Arms: Ubiquinol
Drug: Placebo — Take oral tablets as directed (2x200 mg for 2 months; 1x200 mg for 4 months) with food each morning- upon waking
  Other Names: Sugar pill, inactive substance
  Arms: Placebo

SUMMARY:
The primary objective of this clinical trial is to determine if treatment with ubiquinol, a form of coenzyme Q10, improves the physical function of men and women Veterans suffering from Gulf War Illness (GWI). The primary outcome measure is a change from baseline on the Short Form Health Survey 36-item (SF-36), with respect to physical functioning and symptoms. Secondary outcome measures include changes from baseline levels on GWI-associated biomarkers in peripheral blood and GWI-associated symptoms of chronic pain, fatigue, insomnia, activity level, and cognitive and mental functioning.

DETAILED DESCRIPTION:
As many as a third of the nearly 700,000 military personnel deployed during Desert Shield and Desert Storm (Aug 2, 1990 to July 31, 1991) in the Kuwaiti Theater of Operations are suffering from Gulf War Illness (GWI), an unexplained chronic illness characterized by multiple symptoms. Gulf War Veterans experienced environmental exposures that are known to be oxidative stressors which contribute to cell injury, resulting in mitochondrial dysfunction Exploratory studies using interventions that support cell functioning and prevent or repair stress mediators suggest a role for these targeted interventions, such as Coenzyme Q10. The goal of this clinical trial is to determine if Coenzyme Q10 is effective in increasing physical functioning for Veterans with Gulf War Illness.

This is a randomized, two group, double blind, placebo controlled, Phase III clinical trial. The treatment group will receive a (2x200 mg for 2 months and 1x200 mg for 4 months) once a day of ubiquinol for 6 months. The placebo group will receive matching placebo (2x200 mg for 2 months and 1x200 mg for 4 months) once a day of ubiquinol for 6 months. The primary outcome measure for this clinical trial is a change from baseline of SF-36, with respect to physical functioning and symptoms. The secondary outcome measures include changes from baseline of peripheral blood levels of biomarkers, and of GWI-associated symptoms of chronic pain, fatigue, sleep issues, and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans who were deployed in 1990 -1991 Gulf War.
* Veterans who currently meet the Kansas Gulf War Study Case Definition for Gulf War Illness.
* Veterans who were in good health based on medical history prior to 1990.
* Veterans whose severity of illness is moderate to severe, evidenced by scoring less than 30 of 100 on the physical domain of SF36.

Exclusion Criteria:

* Veteran has a condition that may interfere with the ability to accurately report symptoms, such as:

  * severe psychiatric problems
  * schizophrenia
  * bipolar disorder
  * major depression with psychotic or melancholic features
  * delusional disorders alcohol or drug dependence requiring hospitalization, or regular illegal drug use or other psychiatric condition requiring inpatient stay in the 6 months prior to study entry.
  * Has dementias of any type
  * Currently does not have exclusionary conditions that could reasonably be responsible for the symptoms in multi-symptom disorders, as determined by Investigator (based on Reeves et al.2003).
  * Is pregnant or breastfeeding or plans to become pregnant within the next 6 months.
* Medical conditions excluded:

  * organ failure
  * defined rheumatologic inflammatory disorders
  * chronic active infections such as HIV, hepatitis B and C, or transplant
  * primary sleep disorders
* Medications that could potentially impact immune function excluded:

  * steroids
  * immune-suppressives
  * nutraceuticals that are formulated to impact mitochondrial function or oxidative stress
  * Biologic response modifiers within 3 months of study entry.
* Current use of Coumadin (given the vitamin K structural similarity of CoQ10)
* Known allergy to CoQ10 and/or inactive ingredients of active and placebo soft gelatin capsules
* Willingness to have 12 weeks of washout of current CoQ10, ubiquinol, or ubiquinone supplements will be required between the screening and baseline visits.
* Common multivitamin preparations will be allowed if taken without change throughout the protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy G Klimas, BS MD, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (4):
- United States (4):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ubiquinol | Placebo
Started | 51 | 49
Completed | 41 | 43
Not Completed | 10 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 7 | 4
Not completed — Ubiquinol group -not deployed to Gulf; Placebo group- ill with COVID | 1 | 1

BASELINE CHARACTERISTICS:
Population: Number of all participants for whom baseline characteristics were measured, in each arm/group and in the entire study population (total).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ubiquinol | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intention-to-treat
  years | 54 (6) | 53 (5) | 54 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 46 | 46 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 41 | 36 | 77
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 27 | 32 | 59
  More than one race | 11 | 3 | 14
  Unknown or Not Reported | 1 | 2 | 3
SF 36 Physical Component Summary (PCS) [Mean (Standard Deviation); unit: units on a scale] — The scale is 1-100. The higher value indicates better physical health. Population: Intention-to-treat
  units on a scale | 55 (23) | 56 (22) | 56 (22)

OUTCOME MEASURES:

1. Primary Outcome: Veterans Short Form 36-Item Health Survey Physical Component Summary
Description: Veterans Health Survey contains 36 items to measure health functioning from the patient's point of view. The scale is 0-100. The higher value indicates better physical health.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change Baseline to 4 Weeks | 1.6 (11.1) | -1.1 (10.1)
  Change Baseline to 8 Weeks | 1.4 (12.7) | 1.1 (10.3)
  Change Baseline to 12 Weeks | 1.5 (15.9) | -1.8 (13.1)
  Change Baseline to 16 Weeks | 2.1 (14.5) | 1.8 (12.4)
  Change Baseline to 20 Weeks | 1.6 (14.7) | 0.7 (14.3)
  Change Baseline to 24 Weeks | 0.7 (12.5) | 0.3 (12.7)

2. Secondary Outcome: Multidimensional Fatigue Inventory (MFI)
Description: MFI asks questions about general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. The Multidimensional Fatigue Inventory score is 0-100. The higher value indicates more fatigue.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change Baseline to 4 Weeks | -0.6 (8.3) | 0.2 (10)
  Change Baseline to 8 Weeks | -1.8 (9.9) | 0.5 (8)
  Change Baseline to 12 Weeks | -1.4 (10) | 3.6 (8.4)
  Change Baseline to 16 Weeks | -3.2 (9.5) | 0.3 (8.1)
  Change Baseline to 20 Weeks | -0.5 (7.5) | 2.5 (9.0)
  Change Baseline to 24 Weeks | -2.3 (9.7) | 0.8 (8.7)

3. Secondary Outcome: Gulf War Illness Health Symptom Checklist
Description: The Gulf War Illness Health Symptoms Checklist asks questions about symptoms related to Gulf War Illness. The linear scale is 0-42. The higher value indicates more symptoms.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, and 28
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 4 weeks | -3.7 (8.8) | -2.0 (6.3)
  Change from baseline to 8 weeks | -3.7 (7.5) | -2.6 (9.4)
  Change from baseline to 12 weeks | -5.8 (10.8) | -2.7 (9.4)
  Change from baseline to 16 weeks | -4.6 (9.5) | -1.6 (6.1)
  Change from baseline to 20 weeks | -6.1 (11.9) | -3.7 (10.3)
  Change from baseline to 24 weeks | -3.8 (8.6) | -3.1 (8.0)
  Change from baseline to 28 weeks | -8.7 (11.5) | -9.4 (13.3)

4. Secondary Outcome: Brief Pain Inventory
Description: The Brief Pain Inventory is a linear scale of pain. The scale is 0-10. The higher value indicates more pain.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 4 weeks | 0 (1.1) | 0 (1.3)
  Change from baseline to 8 weeks | -0.1 (1.6) | 0.3 (1.6)
  Change from baseline to 12 weeks | 0.3 (1.7) | 0.3 (1.6)
  Change from baseline to 16 weeks | -0.1 (1.8) | 0.1 (1.4)
  Change from baseline to 20 weeks | 0.2 (1.6) | 0.6 (1.8)
  Change from baseline to 24 weeks | -0.3 (1.4) | -0.3 (1.5)

5. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: The PSQI measures quality and patterns of sleep and wake cycles and is completed by the participant. The Pittsburgh Sleep Quality Index scale is 0-21. The higher value indicates more sleep disturbance.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 4 weeks | -1.0 (2.8) | 0.0 (3.1)
  Change from baseline to 8 weeks | -1.2 (2.9) | -0.4 (2.8)
  Change from baseline to 12 weeks | -1.7 (3.4) | 0.1 (3.6)
  Change from baseline to 16 weeks | -1.6 (3.0) | -1.0 (3.0)
  Change from baseline to 20 weeks | -0.3 (3.7) | 0.3 (3.7)
  Change from baseline to 24 weeks | -1.4 (3.5) | -0.4 (3.5)

6. Secondary Outcome: Hamilton Anxiety Scale (HAM-A)
Description: This measure allows the participant to rate levels of anxiety. The Hamilton Anxiety Scale is 0-56. The higher value indicates more anxiety.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 8 weeks | -0.9 (9.3) | 1.7 (10.3)
  Change from baseline to 16 weeks | -0.7 (8.3) | -1.7 (8.3)
  Change from baseline to 24 weeks | -1.5 (9.0) | 0.1 (10.3)

7. Secondary Outcome: Hamilton Depression Scale (HAM-D)
Description: This measure allows the participant to rate level of depression. The Hamilton Depression Scale is a linear scale 0-62. The higher value indicates more depression.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 8 weeks | -2.4 (6.1) | -1.3 (4.9)
  Change from baseline to 16 weeks | -2.8 (5.8) | -3.6 (4.5)
  Change from baseline to 24 weeks | -2.5 (7.0) | -2.8 (5.8)

8. Secondary Outcome: Veterans Short Form 36-Item Health Survey: Mental Component Score (MCS)
Description: Veterans Health Survey contains 36 items to measure health functioning from the patient's point of view. The Veterans Short Form 36-item Health Survey Mental Component Score scale is 0-100. The higher value indicates more favorable mental health.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 4 weeks | 4.5 (12.6) | 0.4 (12.8)
  Change from baseline to 8 weeks | 4.2 (14.9) | 3.6 (14.8)
  Change from baseline to 12 weeks | 4.0 (19.5) | 2.8 (10.6)
  Change from baseline to 16 weeks | 3.8 (15.5) | 4.9 (13.9)
  Change from baseline to 20 weeks | -3.7 (17.4) | 3.1 (15.8)
  Change from baseline to 24 weeks | 2.6 (16.3) | 1.1 (13.5)

9. Secondary Outcome: Connors Continuous Performance Test (CPT-3): Hit Reaction Time
Description: CPT-3 asks questions about cognitive symptoms related to attention and reaction time. The Connors Continuous Performance Test Hit Reaction Time scale is 0-No limit. The higher score indicates poorer outcomes.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 8 weeks | 10.7 (43.1) | -1.6 (34.3)
  Change from baseline to 16 weeks | 17.2 (46.9) | -3.0 (49)
  Change from baseline to 24 weeks | 24.0 (46.9) | 12.8 (45.4)

10. Secondary Outcome: Connors Continuous Performance Test (CPT-3):Omissions T-score
Description: CPT-3 asks questions about cognitive symptoms related to attention and reaction time. The Connors Continuous Performance Test Omissions score is 0-100. 50 indicates the population mean with a standard deviation of 10. The higher T-score indicates poorer outcomes.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
T-score
  Change from baseline to 8 weeks | -2.0 (7.6) | -1.2 (5.2)
  Change from baseline to 16 weeks | 0.2 (9.1) | -1.6 (8.5)
  Change from baseline to 24 weeks | -0.4 (9.1) | -1.6 (7.8)

11. Secondary Outcome: Connors Continuous Performance Test (CPT-3):Commissions T-score
Description: CPT-3 asks questions about cognitive symptoms related to attention and reaction time. The Connors Continuous Performance Test Commissions T-score scale is 0-100. 50 indicates the population mean with a standard deviation of 10. The higher score indicates poorer outcomes.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
T-score
  Change from baseline to 8 weeks | -3.2 (8.0) | -2.0 (5.3)
  Change from baseline to 16 weeks | -3.2 (8.6) | -3.0 (6.7)
  Change from baseline to 24 weeks | -3.5 (8.8) | -4.5 (7.2)

12. Secondary Outcome: Brief Visual Memory Test (BVMT): Delayed Recall
Description: BVMT asks questions about cognitive symptoms related to visual memory. The Brief Visual Memory Test Delayed Recall scale is 0-12. The higher value indicates better performance.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to8 weeks | 0.3 (2.3) | 0.3 (2.4)
  Change from baseline to 16 weeks | 0.3 (2.8) | 0.9 (2.0)
  Change from baseline to 24 weeks | 0.4 (2.7) | 0.4 (2.2)

13. Secondary Outcome: Brief Visual Memory Test (BVMT): Percent Retained
Description: BVMT asks questions about cognitive symptoms related to visual memory. The Brief Visual Memory Test Percent Retained score is 0-100. The higher value indicates better performance.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 8 weeks | -4.1 (42.9) | 13.7 (43)
  Change from baseline to 16 weeks | -5.6 (24.6) | 1.1 (24.7)
  Change from baseline to 24 weeks | -0.4 (52.3) | 0.4 (39.4)

14. Secondary Outcome: California Verbal Learning Test (CVLT-II): Correct Trials # 1-5
Description: CVLT-II asks questions about cognitive symptoms related to recall and memory. The California Verbal Learning Test (CVLT-II) Correct Trials #1-5 score is 0-80. The higher score indicates better performance.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 8 weeks | 0.4 (7.0) | 0.9 (9.8)
  Change from baseline to 16 weeks | 4.0 (8.4) | 6.7 (7.5)
  Change from baseline to 24 weeks | 5.8 (8.8) | 6.9 (10.0)

15. Secondary Outcome: California Verbal Learning Test (CVLT-II): Short Delay
Description: CVLT-II asks questions about cognitive symptoms related to recall and memory. The California Verbal Learning Test (CVLT-II) Short Delay Test scale is 0-16. The higher score indicates better performance.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
units on a scale
  Change from baseline to 8 weeks | 0.2 (3.0) | 0.5 (2.4)
  Change from baseline to 16 weeks | 1.1 (2.5) | 1.5 (1.9)
  Change from baseline to 24 weeks | 1.1 (2.6) | 1.5 (2.8)

16. Secondary Outcome: California Verbal Learning Test (CVLT-II): Long Delay Test
Description: CVLT-II asks questions about cognitive symptoms related to recall and memory. The California Verbal Learning Test (CVLT-II) Long Delay Test scale is 0-16. The higher score indicates better performance.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 8 weeks | -0.4 (3.7) | 0.6 (2.7)
  Change from baseline to 16 weeks | 0.3 (3.6) | 1.6 (2.8)
  Change from baseline to 24 weeks | 0.9 (2.9) | 1.4 (2.7)

17. Secondary Outcome: Davidson Trauma Scale
Description: Davidson Trauma Scale asks questions about stress, arousal, and avoidance. The scale is 0 - 136. The higher value indicates worse outcome.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
score on a scale
  Change from baseline to 8 weeks | -7.6 (24.6) | -6.7 (23.4)
  Change from baseline to 16 weeks | -5.4 (24.0) | -12.1 (26.5)
  Change from baseline to 24 weeks | -13.3 (18.9) | -9.4 (21.8)

18. Secondary Outcome: FitBit Sleep Measurement - Total Sleep
Description: FitBit measures the duration of sleep daily via a bracelet-type instrument worn on the participant's wrist throughout the study. No normative data for FitBit Sleep was available.
Time Frame: Baseline to 8 weeks, 8 weeks to 16 weeks, 16 weeks to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
minutes
  Average Total Sleep, Baseline to Week 8 | 344.14 (54.6) | 343.4 (59.8)
  Average Total Sleep, Week 8 to Week 16 | 346.31 (60.85) | 348.15 (57.57)
  Average Total Sleep, Week 16 to Week 24 | 350.98 (58.28) | 334.22 (70.86)

19. Secondary Outcome: FitBit Sleep Measurement - Types of Sleep
Description: FitBit measures the time spent in each type of sleep (Light, Deep, Rapid Eye Movement (REM)) daily via a bracelet-type instrument worn on the participant's wrist throughout the study. No normative data for FitBit Sleep was available.
Time Frame: Baseline to 8 weeks, 8 weeks to 16 weeks, 16 weeks to 24 weeks
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: average percentage of total time in bed
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
average percentage of total time in bed
  Asleep, Baseline to Week 8 | 89.06 (2.61) | 88.57 (1.4)
  Asleep, Week 8 to Week 16 | 89.1 (2.6) | 88.5 (1.36)
  Asleep, Week 16 to Week 24 | 88.81 (3.48) | 88.85 (2.06)
  Awake, Baseline to Week 8 | 10.68 (2.71) | 11.34 (1.37)
  Awake, Week 8 to Week 16 | 10.64 (4.28) | 11.43 (1.92)
  Awake, Week 16 to Week 24 | 10.92 (3.28) | 11.09 (2.06)
  Light Sleep, Baseline to Week 8 | 65.37 (6.23) | 64.68 (7.21)
  Light Sleep, Week 8 to Week 16 | 67.31 (6.43) | 65.89 (7.1)
  Light Sleep, Week 16 to Week 24 | 64.49 (6.04) | 65.28 (7.98)
  Deep Sleep, Baseline to Week 8 | 15.29 (3.62) | 14.7 (5.97)
  Deep Sleep, Week 8 to Week 16 | 14.04 (3.97) | 13.82 (5.48)
  Deep Sleep, Week 16 to Week 24 | 15.78 (3.57) | 15.23 (5.86)
  REM Sleep, Baseline to Week 8 | 19.33 (3.86) | 6.41 (1.31)
  REM Sleep, Week 8 to Week 16 | 18.65 (4.38) | 20.21 (3.43)
  REM Sleep, Week 16 to Week 24 | 19.74 (3.98) | 18.75 (4.59)

20. Secondary Outcome: Response to Therapy of Gulf War Illness-associated Peripheral Blood Biomarkers - Complete Blood Count (CBC) White Blood Cell Counts and Platelets
Description: Peripheral blood biomarker levels are quantified by complete blood count (CBC) analyses: white blood cell (WBC) counts and platelets. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: 1000 cells per microliter
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
1000 cells per microliter
  WBC, Change from baseline to 8 weeks | 0.41 (2.63) | 0.34 (1.27)
  WBC, Change from baseline to 16 weeks | 0.22 (2.54) | 0.14 (1.27)
  WBC, Change from baseline to 24 weeks | 0.22 (2.81) | 0.44 (1.44)
  Platelets, Change from baseline to 8 weeks | -0.94 (74.64) | -2.00 (26.20)
  Platelets, Change from baseline to 16 weeks | -5.88 (79.94) | 3.74 (31.36)
  Platelets, Change from baseline to 24 weeks | -6.00 (78.07) | 14.48 (48.81)

21. Secondary Outcome: Response to Therapy of Gulf War Illness-associated Peripheral Blood Biomarkers - Complete Blood Count (CBC) Red Blood Cell (RBC) Counts
Description: Peripheral blood biomarker levels are quantified by complete blood count (CBC) analyses: red blood cell counts. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: 1000000 cells per microliter
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
1000000 cells per microliter
  RBC, Change from baseline to 8 weeks | 0.10 (0.64) | 0.01 (0.27)
  RBC, Change from baseline to 16 weeks | 0.12 (0.70) | -0.03 (0.33)
  RBC, Change from baseline to 24 weeks | 0.08 (0.69) | -0.02 (0.32)

22. Secondary Outcome: Response to Therapy of Gulf War Illness-associated Peripheral Blood Biomarkers - Complete Blood Count (CBC) White Blood Cell Percentages
Description: Peripheral blood biomarker levels are quantified by complete blood count (CBC) analyses: percentages of white blood cells. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
percentage of white blood cells
  Neutrophils, Change from baseline to 8 weeks | 2.08 (15.11) | 1.13 (9.25)
  Neutrophils, Change from baseline to 16 weeks | 0.26 (13.97) | 0.74 (9.36)
  Neutrophils, Change from baseline to 24 weeks | 3.33 (14.81) | 2.04 (10.95)
  Lymphocytes, Change from baseline to 8 weeks | -1.64 (12.29) | -0.39 (7.83)
  Lymphocytes, Change from baseline to 16 weeks | -0.18 (12.73) | 0.10 (7.66)
  Lymphocytes, Change from baseline to 24 weeks | -3.01 (13.22) | -1.01 (8.68)
  Monocytes, Change from baseline to 8 weeks | -0.19 (3.68) | -0.37 (2.36)
  Monocytes, Change from baseline to 16 weeks | -0.43 (2.81) | -0.12 (1.61)
  Monocytes, Change from baseline to 24 weeks | -0.23 (2.88) | -0.39 (1.95)
  Eosinophils, Change from baseline to 8 weeks | -0.25 (2.86) | -0.30 (1.35)
  Eosinophils, Change from baseline to 16 weeks | 0.07 (2.56) | -0.82 (1.86)
  Eosinophils, Change from baseline to 24 weeks | -0.16 (2.67) | -0.67 (2.13)
  Basophils, Change from baseline to 8 weeks | -0.02 (0.69) | -0.06 (0.75)
  Basophils, Change from baseline to 16 weeks | 0.23 (0.54) | 0.14 (0.64)
  Basophils, Change from baseline to 24 weeks | 0.00 (0.64) | 0.07 (0.87)

23. Secondary Outcome: Response to Therapy of Gulf War Illness-associated Peripheral Blood Biomarkers - Complete Blood Count (CBC) Hemoglobin
Description: Peripheral blood biomarker levels are quantified by complete blood count (CBC) analyses: hemoglobin. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
grams per deciliter
  Change from baseline to 8 weeks | 0.18 (1.56) | 0.05 (0.80)
  Change from baseline to 16 weeks | 0.17 (1.59) | -0.25 (0.91)
  Change from baseline to 24 weeks | 0.10 (1.52) | -0.28 (1.11)

24. Secondary Outcome: Response to Therapy of Gulf War Illness-associated Peripheral Blood Biomarkers - Complete Blood Count (CBC) Hematocrit
Description: Peripheral blood biomarker levels are quantified by complete blood count (CBC) analyses: percentages of hematocrit in blood. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
percentage of red blood cells in blood
  Change from baseline to 8 weeks | 0.73 (4.64) | 0.11 (2.58)
  Change from baseline to 16 weeks | 0.63 (4.94) | -0.27 (3.41)
  Change from baseline to 24 weeks | 0.53 (4.77) | -0.25 (3.08)

25. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Thyroid (HPT) Axis: TSH
Description: Thyroid status is assessed using a chemiluminescent method: thyroid stimulating hormone (TSH). Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
mIU/L
  Change from Baseline to Week 8 | 0.344 (1.26) | 0.09 (0.96)
  Change from Baseline to Week 16 | 0.15 (1.31) | -0.06 (0.68)
  Change from Baseline to Week 24 | -0.10 (1.23) | -0.04 (0.92)

26. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Thyroid (HPT) Axis: FT3
Description: Thyroid status is assessed using a chemiluminescent method: Free triiodothyronine (FT3). Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
pg/mL
  Change from Baseline to Week 8 | -0.06 (0.48) | -0.04 (0.29)
  Change from Baseline to Week 16 | -0.13 (0.48) | -0.10 (0.32)
  Change from Baseline to Week 24 | -0.05 (0.56) | -0.17 (0.40)

27. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Thyroid (HPT) Axis: FT4
Description: Thyroid status is assessed using a chemiluminescent method: Free thyroxine (FT4). Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
ng/dL
  Change from Baseline to Week 8 | -0.00 (0.21) | -0.03 (0.11)
  Change from Baseline to Week 16 | -0.01 (0.19) | -0.02 (0.10)
  Change from Baseline to Week 24 | -0.02 (0.18) | -0.06 (0.12)

28. Secondary Outcome: Response to Therapy on Cortisol Levels
Description: Cortisol will be measured using a 24-hour salivary collection to assess circadian rhythm.
Time Frame: Baseline, Weeks 8, 16, and 24 upon waking, mid-morning, evening, and sleep for each.
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
micrograms/dL
  Waking, Change from Baseline to Week 8 | -0.04 (0.32) | -0.04 (0.28)
  Morning, Change from Baseline to Week 8 | 0.04 (0.10) | 0.10 (0.49)
  Evening, Change from Baseline to Week 8 | -0.02 (0.15) | 0.05 (0.19)
  Sleep, Change from Baseline to Week 8 | 0.03 (0.17) | 0.05 (0.23)
  Waking, Change from Baseline to Week 16 | 0.08 (0.63) | 0.02 (0.29)
  Morning, Change from Baseline to Week 16 | 0.12 (0.53) | -0.02 (0.09)
  Evening, Change from Baseline to Week 16 | 0.03 (0.21) | 0.05 (0.21)
  Sleep, Change from Baseline to Week 16 | 0.11 (0.21) | 0.01 (0.13)
  Waking, Change from Baseline to Week 24 | 0.06 (0.24) | 0.03 (0.17)
  Morning, Change from Baseline to Week 24 | 0.02 (0.16) | 0.03 (0.12)
  Evening, Change from Baseline to Week 24 | -0.01 (0.16) | 0.00 (0.12)
  Sleep, Change from Baseline to Week 24 | 0.01 (0.15) | -0.02 (0.11)

29. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Gonadal (HPG) Axis: Testosterone
Description: HPG will measure testosterone. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
ng/mL
  Change from Baseline to Week 8 | -0.12 (2.04) | -0.14 (0.95)
  Change from Baseline to Week 16 | -0.19 (1.99) | -0.39 (0.75)
  Change from Baseline to Week 24 | -0.13 (2.08) | -0.53 (1.30)

30. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Gonadal (HPG) Axis: Progesterone
Description: HPG will measure progesterone. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
ng/mL
  Change from Baseline to Week 8 | 0.01 (0.16) | 0.00 (0.09)
  Change from Baseline to Week 16 | -0.00 (0.16) | -0.03 (0.08)
  Change from Baseline to Week 24 | -0.02 (0.13) | -0.05 (0.06)

31. Secondary Outcome: Response to Therapy on Hypothalamic-Pituitary-Gonadal (HPG) Axis: Estradiol
Description: HPG will measure estradiol. Average values fell within the normal range for this type of assay.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 51 | 49
pg/mL
  Change from Baseline to Week 8 | 6.06 (25.64) | 1.77 (7.51)
  Change from Baseline to Week 16 | -0.97 (11.86) | -1.37 (6.55)
  Change from Baseline to Week 24 | 6.21 (27.90) | -2.19 (8.79)

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: All participants assigned to a study arm or comparison group comprised the at risk population.
Arm/Group | Ubiquinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49

LIMITATIONS AND CAVEATS:
Study recruitment closed on 4/1/2020, coinciding with the onset of the COVID-19 pandemic. Participants could not complete their in-person visits due to the closure of VA research services and VA outpatient labs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02865460/Prot_SAP_000.pdf